CLINICAL TRIAL: NCT00878059
Title: Proxy Decision Making for Alzheimer Disease Research
Brief Title: Alzheimer's Family Research
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: AD R01
Record Dates: First submitted 2009-03-16; First posted 2009-04-08 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Decision Making

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proxies: A family member-caregiver (the medical decision-maker) for someone with Alzheimer's Disease. Must be the person who would be able to make decisions for someone with Alzheimer's disease about being in medical research.

SUMMARY:
This is a research study about how family members make research participation decisions for a relative with Alzheimer's or a related dementia. The purpose of this study is to learn more about how proxies (the family member who makes decisions for that relative), would think through decisions about whether to enroll their relative in studies for not-yet-approved medications for Alzheimer's Disease. The long-term goal of the study is to improve the way researchers inform families about clinical research studies and opportunities for participation. This study is being sponsored by the National Institute on Aging.

Study participants will be interviewed by a research staff member about research enrollment decisions for their relative. A number of standardized questionnaires will be administered. There is only one visit required. The interview lasts about three hours. The investigators will try to make it as convenient as possible for your schedule.

This is a non-intervention study. UCSF CHR # H58055-31168-02 v.1 Date: 012709

DETAILED DESCRIPTION:
* The researcher will interview you for about 3 hours in a private office.
* Study location: All these procedures will be done at Dr. Dunn's research offices at UCSF. If you prefer, we can conduct the interview at your home in or near the San Francisco bay area.
* You will be asked questions about your general background, and about how providing care for the person with Alzheimer's Disease has affected you. You will also be asked some basic questions about the person with Alzheimer's Disease (such as how well they are functioning; personal information will not be collected, however).
* Then, you will be given a consent form for an imaginary study related to Alzheimer Disease. An imaginary study means that it is not a real study, but it is a made-up one. You or your relative will not really participate in the study that is described in the consent form, because it is only imaginary and created just for this research.
* Then, you will be asked questions to measure how well you understood the information presented to you. For example, you will be asked about the procedures, risks and benefits.
* You will also be interviewed regarding your opinions and attitudes about research participation. If you give your permission, we will audiotape this interview to help us more accurately record this information. You may refuse to answer any of the questions that make you uncomfortable. You do not have to agree to be audio-taped to participate in this study.
* You will be given some tests designed to measure memory, attention and other thinking abilities. These tests are for research purposes only, and are not being used for any type of diagnostic purposes. The research purpose is to help us understand proxies' abilities to make decisions as caregivers for seriously ill patients.
* You will be asked questions about your mood and about caring for someone with dementia. You may refuse to answer and questions that make you uncomfortable.

ELIGIBILITY:
Inclusion Criteria:

* A family member-caregiver (the medical decision-maker) for someone with Alzheimer's Disease
* Able to be interviewed in person in or around the San Francisco Bay Area
* Able to read and understand English

Exclusion Criteria:

* People who do not meet inclusion criteria or who become uncooperative or unwilling to complete the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be adult men and women who, under California law (AB2328), would be legally eligible to serve as proxy decision makers for Alzheimer's Disease patients for research. These will be spouses or adult children of people with Alzheimer's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura B Dunn, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Langley Porter Institute, or at participant's home, San Francisco, California, United States